CLINICAL TRIAL: NCT07407478
Title: Effect of Foot Core Exercises on Jump Performance in Professional Volleyball Players: An Objective Evaluation Using ForceDecks
Brief Title: Effect of Foot Core Exercises on Jump Performance in Professional Volleyball Players
Acronym: FCJUMP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mudanya University (Other)
Responsible Party: Principal Investigator, Hazal Berfin YILMAZ, Study Director, Mudanya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025/222
Record Dates: First submitted 2026-01-03; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Athletic Performance
Keywords: Foot Core Exercise; Jump Performance; Volleyball Players; Countermovement Jump; Force Plates; Athletic Performance

STUDY DESIGN:
Intervention Model Description: This study is designed using a parallel assignment model. Participants will be randomly allocated into two groups. The first group will perform a standardized strength training program only, while the second group will perform foot core exercises in addition to the same strength training program. Both groups will be followed simultaneously throughout the intervention period.
Masking Description: This study is conducted as an open-label trial. Both participants and researchers are aware of the interventions being administered. There are no additional parties masked in this clinical study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength Training Group (Active Comparator): Description Participants in this group will perform a standardized lower-extremity strength training program routinely used for professional volleyball players.
  Interventions: Behavioral: Strength Training Program
- Strength Training plus Foot Core Exercise Group (Experimental): Experimental: Strength Training Plus Foot Core Exercises Group
  Description Participants in this group will perform the same standardized lower-extremity strength training program in addition to a foot core exercise program targeting intrinsic and extrinsic foot muscles.
  Interventions: Behavioral: Strength Training Program; Behavioral: Foot Core Exercise Program

INTERVENTIONS:
Behavioral: Strength Training Program — Description Participants will perform a standardized lower-extremity strength training program routinely used for professional volleyball players.
  Arms Assigned
  * Strength Training Group
  * Strength Training Plus Foot Core Exercises Group
Behavioral: Foot Core Exercise Program — Description Participants will perform foot core exercises targeting intrinsic and extrinsic foot muscles. The exercises are designed to improve foot stability and functional control.
  Arms Assigned ✔️ Strength Training Plus Foot Core Exercises Group
  ❌ Strength Training Group (işaretleme)
  Arms: Strength Training plus Foot Core Exercise Group

SUMMARY:
Brief Summary

The purpose of this study is to investigate the effect of foot core exercises on jump performance in professional volleyball players. Participants will be randomly assigned to two groups. The first group will perform a strength training program only, while the second group will perform foot core exercises in addition to the same strength training program. Jump performance will be assessed using the Countermovement Jump (CMJ) test, and performance scores will be obtained through force-time analysis using the ForceDecks system. The findings of this study are expected to contribute to the development of training programs aimed at improving performance and reducing injury risk in professional volleyball players.

DETAILED DESCRIPTION:
Detailed Description

This study is designed to examine the effects of foot core exercises on jump performance in professional volleyball players. Participants will be divided into two groups: a control group and an intervention group. The control group will follow a standardized strength training program, while the intervention group will perform the same strength training program combined with additional foot core exercises.

Jump performance will be evaluated using the Countermovement Jump (CMJ) test. Kinetic variables derived from force-time data will be collected using the ForceDecks system. Pre- and post-intervention measurements will be compared to determine the effects of the training programs.

The results of this study are expected to provide evidence-based information for designing training programs that enhance athletic performance and help reduce injury risk in professional volleyball players.

ELIGIBILITY:
Inclusion Criteria:

* Male professional volleyball players aged 18 to 35 years
* Actively licensed athletes competing in clubs affiliated with the Turkish Volleyball Federation
* Regular participation in team training sessions without interruption for at least the past 3 months
* No history of surgery or serious injury involving the lower extremities (foot, ankle, knee, or hip) within the last 6 months
* Agreement not to participate in any additional strength, balance, or proprioception-based exercise programs during the study period
* No medical or physiological condition that would prevent participation in the Countermovement Jump (CMJ) test performed using the ForceDecks system
* Voluntary participation with written informed consent obtained prior to enrollment

Exclusion Criteria:

* Presence of deformity, chronic pain, or functional impairment in the foot or ankle
* History of lower extremity orthopedic surgery within the past 6 months
* History of neurological or vestibular disorders, or systemic diseases affecting balance
* Participation in physiotherapy interventions, rehabilitation protocols, or exercise programs outside the scope of the study during the study period

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male professional volleyball players are eligible to participate in this study.
Enrollment: 43 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Vertical Jump Height (Countermovement Jump) | Baseline and post-intervention (approximately 8 weeks)
  Maximum vertical jump height measured during the Countermovement Jump (CMJ) test.

SECONDARY OUTCOMES:
Force-Time Variables During Countermovement Jump | Baseline and post-intervention (approximately 8 weeks)
  Force-time variables obtained from force platform measurements during the Countermovement Jump (CMJ) test.

CONTACTS AND LOCATIONS:
Overall Officials: Hazal B Yılmaz, PhD, Principal Investigator — Mudanya University
Locations (1):
- Mudanya University, Bursa, Mudanya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, as this study is conducted as part of a master's thesis with a limited sample size, and data sharing is not covered by the informed consent approved by the ethics committee.